CLINICAL TRIAL: NCT00803894
Title: A Randomized Clinical Trial to Study the Effects of MK0752 Versus Placebo on Biomarkers in Healthy Young Adult Male Subjects
Brief Title: A Clinical Study to Determine Biomarkers of Response to a Gamma Secretase Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0752-022; 2008_594
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Biomarkers of Notch inhibition
MeSH Terms: interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): MK0752 1000 mg
  Interventions: Drug: MK0752
- B (Active Comparator): MK0752 350 mg
  Interventions: Drug: Comparator: MK0752.
- C (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK0752 — Single dose MK0752 capsules, 1000 mg: there will be a 7-day washout period between treatments.
  Arms: A
Drug: Comparator: MK0752. — Single dose MK0752 capsules, 350 mg: there will be a 7-day washout period between treatments.
  Other Names: MK0752
  Arms: B
Drug: Comparator: Placebo — Single dose placebo capsules: there will be a 7-day washout period between treatments.
  Arms: C

SUMMARY:
The purpose of this study is to determine the transcriptional signature of Notch Inhibition by testing hair and blood samples on healthy male volunteers who have received MK0752 vs placebo for possible future biomarkers in the treatment of cancer or Alzheimers Disease

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male
* Patient has no clinically significant abnormality on electrocardiogram performed
* Patient agrees to not to consume apple juice, grapefruit or grapefruit products beginning 2 weeks prior to first dose of study drug and for the duration of the study
* Patient has been a nonsmoker and/or has not used nicotine or nicotine-containing products for approximately 6 months.
* Patient is willing to not use any hair enhancement product or procedures for the duration of the study (for example, permanents, hair straightening techniques)
* Patient has a full head of hair
* Patient has at least 90% non-gray hair

Exclusion Criteria:

* Patient has had treatment with any investigational therapy during the prior 21 days
* Patient has any history of significant gastrointestinal abnormalities within the last 10 years
* Patient has a history of any long-term or active liver disease including elevated liver blood tests. Any patient with a history of Hepatitis B or C (and/or treated previously) will be excluded
* Patient has a known history or family history of aortic valve disease, congenital (from birth) heart disease or deafness, hearing loss or early onset Alzheimer's disease (onset at age < 55)
* Patient has a known sensitivity to the ingredients in the drug
* Patient has had active and uncontrolled infection within the past month
* Patient is HIV positive
* Patient has a history of stomach, intestine, heart, blood, liver, brain, kidney, lung, bladder or endocrine abnormalities or diseases
* Patient has a history of cancer except for certain skin cancer (basal cell)
* Patient has a history of multiple and/or severe allergies or has had an allergic reaction to food or prescription/non-prescription drugs
* Patient has had major surgery, donated or lost 1 unit of blood (about 500 mL) within the past month
* Patient has premature graying hair (> 10% gray hair)
* Patient has male pattern hair loss
* Patient has a prior history of high blood pressure
* Patient uses any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort) beginning approximately 2 weeks prior to the first dose of study drug, throughout the study until the post study visit
* Patient consumes excessive amounts of alcohol (greater than 3 glasses of alcoholic beverages)
* Patient consumes excessive amounts (greater than 6 servings) of coffee, tea, cola or other caffeinated beverages per day
* Patient is a regular use (including "recreational use") of any illicit drugs, has a positive urine drug screen before randomization or has a history of drug (including alcohol) abuse within approximately the past 2 years
* Patient has prior exposure to MK 0752 with the past 21 days

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the existing Notch response signature using plucked hair follicle profiling data from health young male volunteers given 1000 mg MK0752 and 350 mg MK0752. | 8.5 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Tanis KQ, Podtelezhnikov AA, Blackman SC, Hing J, Railkar RA, Lunceford J, Klappenbach JA, Wei B, Harman A, Camargo LM, Shah S, Finney EM, Hardwick JS, Loboda A, Watters J, Bergstrom DA, Demuth T, Herman GA, Strack PR, Iannone R. An accessible pharmacodynamic transcriptional biomarker for notch target engagement. Clin Pharmacol Ther. 2016 Apr;99(4):370-80. doi: 10.1002/cpt.335. Epub 2016 Feb 17. PMID 26765077